CLINICAL TRIAL: NCT03286907
Title: A Randomized Controlled Trial Evaluating Efficacy of Promoting Human Papillomavirus (HPV) Vaccination Among Chinese Men Who Have Sex With Men
Brief Title: An RCT Promoting HPV Vaccination Among Chinese MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMRF13141651
Record Dates: First submitted 2017-08-28; First posted 2017-09-19 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Health Behavior
Keywords: Uptake of HPV vaccination
MeSH Terms: conditions — Health Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online videos (Experimental): Participants will watch two online videos, complete a self-administered online tutorial, and receive reminders at Month 1, 2, 4, 6 & 8
  Interventions: Behavioral: Online videos
- Online videos and MI (Experimental): Participants will watch two online videos, complete a self-administered online tutorial, received motivational interviewing (MI), and receive reminders at Month 1, 2, 4, 6 & 8
  Interventions: Behavioral: Online videos and MI
- Control group (Active Comparator): Participants will receive online messages about mental health problems and stress reduction exercises
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Online videos — Watch two online short health promotion videos (five minutes each), complete a self-administered online exercise and receive reminders at month 1, 2, 4, 6 & 8.
  Arms: Online videos
Behavioral: Online videos and MI — Watch two online short health promotion videos (five minutes each), complete a self-administered online exercise, receive 15 minutes motivational interviewing through telephone and reminders at month 1, 2, 4, 6, & 8.
  Arms: Online videos and MI
Behavioral: Control group — Receive online health communication messages about prevalence of some common mental health problems among MSM and introduction of stress reduction exercises
  Arms: Control group

SUMMARY:
Objectives:

To evaluate efficacies of two online and theory-based interventions [HC: health communication only and HC-MI health communication plus motivational interviewing (MI)] in increasing uptake of three doses of HPV vaccines within the 9-month follow-up period among Hong Kong Chinese men who have sex with men (MSM).

Hypothesis:

The HPV vaccination rate of the three groups would be in the order HC-MI group > HC group > Control group.

Design and subjects:

A three-arm randomized controlled trial (RCT) will be conducted (n= 624). With informed consent, anonymous surveys will be conducted at baseline, Months 3, 6, and 9. Inclusion criteria: 1) HK Chinese men aged >18, 2) oral or anal intercourse with men in the last six months; 3) no intention to leave HK for one month consecutively within the next 12 months, 4) regular internet access, and 5) willing to be followed up by phone.

Study instruments:

Structured questionnaires

Interventions:

1) Group HC: exposure to web-based, interactive and theory-based health communication promoting HPV vaccination uptake; 2) Group HC-MI: same exposure as Group HC plus MI; and 3) Group C: exposure to online materials about mental health (control group).

Main outcome measures:

Uptake of three doses of HPV vaccination within the follow-up period.

Data analysis and expected results:

Intention-to-treat analysis, General Estimation Equation (GEE) and Cox regression methods will be used. Significance differences in HPV vaccination uptake rates will be found among the three groups.

DETAILED DESCRIPTION:
Aims and objectives

1. The primary objective of the RCT study is to evaluate the relative efficacies of two online, theory-based and interactive interventions [health communication (HC) and health communication plus MI (HC-MI)] in increasing uptake of three required doses of HPV vaccination within a 9-month follow-up period among Hong Kong Chinese MSM who had not previously taken up any dose of HPV vaccination, as compared to the control group (Group C)
2. Secondary objectives are to evaluate the relative efficacies of the interventions in increasing the following responses at the end of the 9-month follow up period:

   i) Intention to take up all doses of HPV vaccination in the next 12 months. ii) Theory-based cognitions supportive of HPV vaccination [e.g. those of the Health Belief Model (HBM)].

   Study design A three-arm parallel RCT will be conducted. Background information and potential confounder(s) are recorded at baseline. Three post-intervention evaluations will be performed through short telephone surveys 3, 6 and 9 months after exposure to the intervention. Participants who have already taken up all three doses of HPV vaccination at Month 3 or 6 will be asked the termination questionnaire (same as that for Month 9). Interviewers and data analysts are blinded from participants' randomization status.

   Subject Inclusion criteria: 1) Hong Kong Chinese speaking men of aged ≥18, 2) self-reported oral or anal intercourse with ≥1 man (last six months); 3) no intention to leave Hong Kong for >1 month consecutively within the next nine months, 4) regular internet access and 5) willing to be followed up by phone. Those who have ever received HPV vaccination will be excluded.

   Recruitment procedures Participants will be recruited by outreaching in local gay-friendly venues. The fieldworkers will explain the study's detail to participants. Verbal instead of written informed consent will be obtained due to the need to maintain anonymity; the fieldworkers will sign a form pledging that participants have been fully briefed and participants' verbal informed consent was obtained. Fieldworkers obtain multiple contacts (mobile, email and/or other e-contact) from prospective participants. Participants will also be recruited via the Internet by comparable procedures.

   Ethical considerations Fieldworkers guarantee anonymity, the right to quit at any time and that refusal will not affect participants' chance in using any services. Verbal instead of written informed consent will be obtained due to the need to maintain anonymity; the fieldworkers will sign a form pledging that participants have been fully briefed. In addition, all participants will reconfirm informed consent online before receiving the online intervention; if the participants select "refuse" for the online informed consent form, the program will close automatically. Ethics approval was obtained from the Survey and Behavioral Research Ethics Committee of the CUHK and the Joint CUHK-NTEC Clinical Research Ethics Committee. All information will be kept in locked areas.

   Randomization In the pre-arranged phone call, fieldworkers brief prospective participants again and reconfirm participants' informed consent. Participants are randomly allocated into one of the three groups, with a sealed opaque envelop drawn by the research staff. Computerized random numbers and block randomization (block size of 12) will be used.

   Primary and secondary outcomes The primary outcome of the study is whether the participant has taken up all three doses of HPV vaccination (at any clinic) within a 9-months follow-up period. Secondary outcomes include intention to take up all three doses of HPV vaccination in the next 12 months and changes in HBM-related cognitions on HPV.

   The baseline survey After randomization takes place, the fieldworker will administer a baseline telephone survey to record information on potential confounders (Questionnaire A: 10-15 minutes).

   Evaluation surveys at Months 3, 6 and 9 A short interim phone interview will be administered at Month 3 and 6 to those who have not taken up three doses of HPV vaccination at Months 3 and 6 (non-termination) after exposure to intervention, recording only uptake of HPV vaccination (one dose or two doses, price, venue and date) during the inter-survey intervals and intention to take up three doses of vaccination in the next 12 months (Questionnaire B, <5 minutes). Participants present at Month 9 or having taken up all three dose at Month 3 and 6 (termination) will be asked about HPV vaccination history, as well as cognitive perceptions and emotional factors included in the baseline survey (Questionnaire C, about 10 minutes). To reduce loss-to-follow-up, the investigators will show these questionnaires to the participants at baseline.

   Information for validating vaccine uptake All participants, including those who are vaccinated at the collaborating clinic, will be requested to send the research team an image of the receipt, hiding personal identification and via the same smartphone number, social media account, or email previous used in this project, after participants have taken up each dose of HPV vaccines.

   Intervention of the Group HC (Online Health Communication Only Group) Participants will watch two short health promotion videos (five minutes each), which contain health communication messages about HPV and HPV vaccination and complete a self-administered exercise which attempts to increase related knowledge and supportive cognitions. After completing the tutorials, participants will be requested to answer an online questionnaire that contains only three simple questions asking about some details of the two videos. This is to verify exposure to the videos. One's login time for the tutorial will be recorded by the computer program (another way to cross-check exposure).

   Intervention of the Group HC-MI (Online Health Communication Plus MI Group) In addition to the components received by the Group HC, Group HC-MI will receive motivational interviewing (MI) of 15 minutes. To increase involvement of the interviewer and rapport, the interviewer will "wait for" the participants while the participants are performing the tutorial. [The interviewer will hold (via third line holding) or hang up the phone while the participant is doing the tutorial and call back 20 minutes afterwards]. The interviewer will discuss briefly about the tutorial (e.g. participants' responses or questions) with the participants to enhance support and also to verify exposure to the tutorial. The interviewer will then conduct a 15-minute MI session with the participant over phone.

   Maintenance of motivation for Group HC and Group HC-MI In order to maintain motivation formed during the intervention, tailored reminders will be sent by Whatsapp or emails to all participants of the Group HC and Group HC-MI. A link to the project webpage will be included in such reminders, prompting participants to access a webpage where participants can watch a testimonial video about HPV experience presented by a peer MSM, read comments made by other participants, add participants' own comments and feedback on others' comments. Such arrangements will provide continuous cues to action for maintaining motivation. The number of reminders will be standardized to five (at month 1, 2, 4, 6 & 8). The number of reminders sending to participants who have taken up all three doses of HPV vaccination will be recorded.

   The control group (Group C) The health communication messages in Group C will consist of online messages about prevalence of some common mental health problems among MSM and introduction of stress reduction exercises. No reminder will be given.

   Sample size planning For planning purpose, the investigators conservatively assume 30% of the automated health communication intervention (Group HC) would show an intention, and 40% of those with such an intention would actually take up HPV vaccination (i.e. 12% of Group HC). Regarding the Group HC-MI, the investigators assume the intention would increase to 60% as MI is a powerful tool; the investigators assume that 50% of its members with an intention would actually take up the vaccine (hence 30% of Group HC-MI would be vaccinated). A sample size of 113 per group is needed to achieve the planned effect sizes and power of .8 and alpha of .0125 for all comparisons (taking into account multiple comparisons). With an expected loss-to-follow up rate of 35% at month 9, a sample size of about 174 per group is required (total n=522). To be conservative, the investigators keep the target sample size of 208 per group (624 in total); which can detect smallest between-group difference of 16.2% between Group HC (12%) and Group HC-MI (~28.2%), and detect smallest between-group difference of 10% between Group HC (12%) and Group C (~2%), at power of .8 and alpha of .0125 (taking into account multiple comparisons).

   Data processing and analysis Test-retest reliability of the baseline questionnaire will be assessed. For categorical responses, Cohen's Kappa statistics will be tested, while for continuous responses, intra-class correlation coefficient will be used. Chi-square test or one-way ANOVA will be conducted to compare differences in background characteristics of those being followed up and loss to follow-up, and differences in potential confounders recorded at baseline among the three groups.

   Intention-to-treat analysis will be performed to assess relative efficacy of the two interventions Generalized Estimation Equation (GEE) models will be fit to investigate significance of differences in primary and secondary outcomes across the three groups, adjusted for any significant potential confounders. Absolute and relative risk reductions and corresponding 95% CI will be derived. Cox regression analysis will also be performed, treating those who are loss to follow-up during the follow-up period and those who had not taken up all three doses of HPV vaccination at the end of the 9-month follow-up period as censored cases, and completion of all three doses of HPV vaccination as the event (endpoint), and intervention group membership as the covariate. Adjustment for potential confounders (found to be significant at baseline analysis) will be performed if necessary.

ELIGIBILITY:
Inclusion Criteria:

* HK Chinese speaking men of aged ≥18
* Self-reported oral or anal intercourse with ≥1 man (last six months)
* No intention to leave HK for >1 month consecutively within the next nine months
* Regular internet access
* Willing to be followed up by phone.

Exclusion Criteria:

* Had ever received HPV vaccination

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Uptake of three required doses of HPV vaccination | 24 months
  Uptake of three required doses of HPV vaccination within a 24-month follow-up period

SECONDARY OUTCOMES:
Behavioral intention to take up all doses of HPV vaccination | 12 months
  "How likely will you take up all three doses of HPV vaccination in the next 12 months?" (Response categories: 1=very unlikely, 4=very likely)

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, PhD, Principal Investigator — Centre for Health Behaviours Research, JC School of Public Health and Primary Care, The Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Wang Z, Lau JTF, Ip TKM, Yu Y, Fong F, Fang Y, Mo PKH. Two Web-Based and Theory-Based Interventions With and Without Brief Motivational Interviewing in the Promotion of Human Papillomavirus Vaccination Among Chinese Men Who Have Sex With Men: Randomized Controlled Trial. J Med Internet Res. 2021 Feb 2;23(2):e21465. doi: 10.2196/21465. PMID 33528372